CLINICAL TRIAL: NCT06897735
Title: A Phase I Pilot Study to Evaluate the Bioequivalence, Pharmacokinetics, and Safety of Inhaled Afatinib Dimaleate Compared to the Reference Oral Afatinib Dimaleate in Healthy Smoking Volunteers (EDDIS-a1)
Brief Title: Exploratory Study of Inhaled Afatinib Dimaleate PK Profile
Acronym: EDDIS-a1
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Petrov, Andrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 233-1-10AfD
Record Dates: First submitted 2025-03-02; First posted 2025-03-27 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer; Oral Cancer; Melanoma
Keywords: Afatinib Dimaleate; BIBW2992 Dimaleate; GIOTRIF; GILOTRIF
MeSH Terms: conditions — Lung Neoplasms; Mouth Neoplasms; Melanoma | interventions — Afatinib

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive inhaled or oral Afatinib Dimaleate treatment first, followed by a washout period, after which they will receive the alternative treatment Participants will receive either a single dose of inhaled afatinib dimaleate or 40 mg of oral afatinib dimaleate in a randomized sequence with a 7-day washout period between treatments.
  Inhaled afatinib dimaleate (liquid) is delivered using a maintenance-free, single-use ultrasonic nebulizer that generates aerosol particles of a defined size with the most efficient gas-dynamic characteristics for alveolar deposition. Each inhalation session consists of a defined number of breaths, which ensures the most efficient uptake of afatinib dimaleate aerosol in the lungs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Afatinib Dimaleate inhalation form (liquid for inhalation) (Experimental): Single-dose administration of inhaled afatinib dimaleate via an ultrasonic inhaler (healthy volunteer smokers only)
  Interventions: Drug: Afatinib Dimaleat; Biological: inhalation of afatinib dimaleate
- Reference Afatinib Dimaleate (Active Comparator): Single oral administration of reference afatinib dimaleate 40 mg capsule (healthy volunteer smokers only)
  Interventions: Drug: Afatinib Dimaleat; Biological: inhalation of afatinib dimaleate

INTERVENTIONS:
Drug: Afatinib Dimaleat — printed capsule containing 40 mg afatinib dimaleate
  Other Names: BIBW2992 Dimaleate; Gilotrif; Afatinib Dimaleate
Biological: inhalation of afatinib dimaleate — inhalation stable form of afatinib dimaleate at an equivalent therapeutic dose in a single-use maintenance-free ultrasonic inhaler with controlled frequency and number of inhalations
  Other Names: Afatinib Dimaleate; BIBW2992 Dimaleate

SUMMARY:
This is a pilot Phase I open-label randomized single-dose two-period crossover study (in the EDDIS project) evaluating the bioequivalence, pharmacokinetics (PK), safety, and tolerability of inhaled afatinib dimaleate compared with the reference oral afatinib dimaleate in healthy volunteer smokers.

The study will enroll healthy adult volunteers smoker to assess the systemic exposure and lung deposition of inhaled afatinib dimaleate. Participants will receive both the test inhaled formulation and the reference oral formulation in separate periods with delayed phase between treatments.

Key endpoints include maximum plasma concentration (Cmax), area under the concentration-time curve (AUC), and lung deposition assessed via bronchoalveolar lavage (BAL), frequency of occurrence of side effects and cases of toxicity during the studies

DETAILED DESCRIPTION:
Participants will receive either a single dose of inhaled afatinib dimaleate or a 40 mg oral dose of afatinib dimaleate in a randomized sequence, with a 7-day washout period between treatments.

The inhaled formulation of afatinib dimaleate is administered via a single-use, maintenance-free ultrasonic nebulizer (by SWITZERLAND TEAM) that generates aerosol particles of a defined size, ensuring predictable bioavailability and targeted alveolar deposition. Each inhalation session consists of a predefined number of physiological breaths, facilitating efficient drug uptake into the lungs at therapeutically relevant doses.

Key assessments include blood sampling for pharmacokinetic (PK), LC-MS/MS, analysis, bronchoalveolar lavage (BAL) to evaluate pulmonary drug deposition, and spirometry to assess pulmonary safety.tests, CT.

The investigators aim to obtain data on the role of pulmonary P-glycoprotein (P-gp) transporters in actively expelling afatinib dimaleate back into the alveolar space, as well as its metabolism by cytochrome P450 enzymes (CYP3A4) during inhalation.

Additionally, statistically significant data on both drug lung deposition (DLD) and drug-induced lung injury (DILI) will be analyzed.

Pharmacokinetic parameters, including maximum plasma concentration (Cmax) and area under the concentration-time curve (AUC0-∞), will be evaluated through plasma sampling. BAL will be performed in a subset of participants to assess direct pulmonary drug deposition. Safety and tolerability will be monitored through adverse event reporting, laboratory testing, and spirometry.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers aged 21 to 55 years
* Body mass index (BMI) from 18.5 to 30.0 kg/m²
* Smokers or people who use e-cigarettes or vapes
* No history of serious lung disease or respiratory disorders
* No history of EGFR-targeted therapy or chemotherapy
* Ability to give informed consent and comply with study procedures

Exclusion Criteria:

* Pregnancy or lactation. (for female participants - 2 negative tests 10 days and 3 days before the start of the study)
* Significant cardiovascular, hepatic, renal or neurological disorders. (ECG 30 days or earlier before the start of the study)
* Recent use of any study drug (within 30 days) or prescription drugs that may affect the metabolism of afatinib
* Known hypersensitivity to afatinib, its salts or derivatives of afatinib or related compounds
* Рarticipation in other studies

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-09 (Estimated); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-05-07 (Estimated)

PRIMARY OUTCOMES:
Cmax (maximum observed plasma concentration) | up to 48 hours post-dose
  quantitative measurement of afatinib dimaleate in plasma
afatinib dimaleate urinary concentrations | up to 96 hours
  quantitative measurement of afatinib dimaleate in urine of inhaled and oral afatinib dimaleate

SECONDARY OUTCOMES:
AUC (Area Under the Plasma Concentration-Time Curve) | up to 48 hours post-dose/inhalations
  the total afatinib dimalete exposure integrated over time

OTHER OUTCOMES:
Determination of afatinib dimaleate concentration in blood | up to 96 hours
  LC-MS/MS (liquid chromatography with selective mass analysis)
Median percentage of total neutrophils relative to absolute neutrophil count | up to 96 hours
  BAL (bronchoalveolar lavage)
  CAUTION! Bronchoalveolar lavage (BAL) should be distinguished from bronchial lavage (when a saline solution is injected into the large airways or bronchi and the fluid is then aspirated for analysis)

CONTACTS AND LOCATIONS:
Locations (1):
- Central Contact, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No